CLINICAL TRIAL: NCT00315887
Title: A Double-Blind Comparative Study of Buprenorphine Transdermal System (BTDS) and Hydrocodone/Acetaminophen Tablets in Patients With Chronic Back Pain
Brief Title: The Safety and Efficacy of the Buprenorphine Transdermal Delivery System in Subjects With Chronic Back Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP98-1201
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-04

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; opioid; transdermal
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Drug: Buprenorphine transdermal delivery system

SUMMARY:
The objective of this study is to assess the safety and efficacy of the buprenorphine transdermal system (5, 10, and 20 mg) in comparison to placebo transdermal system and hydrocodone/acetaminophen in subjects with chronic back pain. The double-blind treatment intervention duration is 56 days during which time supplemental analgesic medication (ibuprofen) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain. Transdermal systems may offer advantages over currently indicated oral products including ease and convenience of use, improved compliance, possible reduction in patient care, and prolonged and consistent delivery of drug.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence of chronic back pain related to intervertebral disc disease, nerve root entrapment, spondylolithesis, osteoarthritis, or other, similar nonmalignant conditions.
* back pain treated with an opioid-containing analgesic at a dose equal to or less than the equivalent of 90 mg of oral morphine per day or 12 or fewer capsules or tablets of an opioid combination analgesic per day.

Exclusion Criteria:

* receiving opioids at an average daily dose of greater than 90 mg of oral morphine equivalents or patients receiving more than 12 tablets per day of short-acting opioid-containing products.
* scheduled to have surgery (including dental) during the study period that involved the use of pre- and/or postoperative analgesics or anesthetics.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 1999-04; Study Completion 1999-10

PRIMARY OUTCOMES:
Patient Satisfaction With Medication for Pain and Average Pain Intensity scores on days 0, 7, 14, 21, 28, 35, 42, 49, 56 and, if applicable, at early termination.

SECONDARY OUTCOMES:
Average Pain Intensity and Patient Satisfaction With Medication for Pain scores (Patient Global Efficacy Rating)
incidence of and time to early discontinuation due to lack of efficacy
investigator's assessment of therapeutic response
dose level at the end of titration

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Arthritis Center of Connecticut, Waterbury, Connecticut
  - University Clinical Research, DeLand, Florida
  - Gainesville Clinical Research Center, Gainesville, Florida
  - Miami Research Associates, Miami, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - Coastal Medical Research, South Daytona Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Private Practice, Weston, Florida
  - Pain Management & Rehabilitation, Terre Haute, Indiana
  - Mid-America Rheumatology Consultants, Overland Park, Kansas
  - Riverhills Healthcare, Crestview Hills, Kentucky
  - Arthritis & Osteoporosis Treatment & Research Center, Jackson, Mississippi
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - PrecisionMed, Inc., Las Vegas, Nevada
  - Cornerstone Research Care, High Point, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Center for Clinical Research, Austin, Texas
  - The Arthritis Clinic of Northern Virginia, Arlington, Virginia
  - Evergreen Clinical Research, Edmonds, Washington
  - Private Practice, Wauwatosa, Wisconsin